CLINICAL TRIAL: NCT01069510
Title: Heart Failure in Congenital Heart Disease: the Role of Myocardial Fibrosis. Treatment Sub-Study: Spironolactone vs. Placebo
Brief Title: Spironolactone in Adult Congenital Heart Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Oregon Clinical and Translational Research Institute (Other)
Responsible Party: Principal Investigator, Craig Broberg, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: eIRB 5845; K23HL093024-01A1 (NIH)
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-07

CONDITIONS: Congenital Heart Disease; Heart Failure; Endomyocardial Fibrosis
MeSH Terms: conditions — Heart Defects, Congenital; Heart Failure; Endomyocardial Fibrosis | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Patients will receive placebo
  Interventions: Other: Placebo
- Spironolactone (Experimental): Spironolactone 25 mg daily
  Interventions: Drug: Spironolactone 25mg

INTERVENTIONS:
Drug: Spironolactone 25mg — Spironolactone 25 mg daily for 12 months
  Other Names: Aldactone 25 mg daily
  Arms: Spironolactone
Other: Placebo — Placebo daily for 12 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if the study drug called spironolactone reduces fibrous (stiffening) in heart muscle tissue and improves heart function. Subjects from the study titled "Heart Failure in Congenital Heart Disease: the role of myocardial fibrosis" who have evidence of heart dysfunction and/or evidence of fibrosis (stiffening) in the heart muscle will be asked to take part in this study.

DETAILED DESCRIPTION:
This study will include randomizing the subject to receive the study drug or placebo. Randomization will occur during visit 1.

Visit 1 will include the following:

* Subjects will answer questions about how well they can breathe.
* An MRI. Dye called gadolinium will be injected into the subject's vein.
* They will go to the Oregon Clinical and Translational Research Institute where 2 tablespoons of blood will be drawn from an intravenous (IV) catheter (tube).
* They will do a 6 minute walk test..
* They will also have an echocardiogram, which is a test that looks at the movement of the subject's heart. A technician will place a cool jelly on their chest and use a small wand to take pictures through the skin.

Subjects' will also have visits 3-6 weeks, 3, 6, 9 months, and 12 months after randomization. Visits 2-5 will include the following:

* They will go to the Oregon Clinical and Translational Research Institute where 1/2 tablespoon of blood will be drawn.
* They will do a 6 minute walk test. During this test, they will walk back and forth in a hallway. The goal is to walk as far as possible for 6 minutes. Subjects will probably get out of breath or become exhausted. If they do, they can slow down, stop, or rest as they need to. Blood pressure will be taken before the walk.
* They will have a health review at 6 months.

Visit 6 will be identical to visit 1 and include the following:

* Subjects will answer questions about how well they can breathe.
* An MRI. Dye called gadolinium will be injected into the subject's vein.
* They will go to the Oregon Clinical and Translational Research Institute where 2 tablespoons of blood will be drawn from an intravenous (IV) catheter (tube).
* They will do a 6 minute walk test..
* They will also have an echocardiogram, which is a test that looks at the movement of the subject's heart. A technician will place a cool jelly on their chest and use a small wand to take pictures through the skin.

The investigators will compare the study drug, called spironolactone, to placebo with regard to any changes in heart stiffening and function of the heart.

ELIGIBILITY:
Inclusion Criteria:

1. Fibrosis index ≥29%, or
2. Evidence of cardiovascular dysfunction including any of the following:

   * Systemic ejection fraction <55%,
   * NYHA 2-3
   * 6-minute walk distance <500 m.
3. Completion of Visit 1 of the study Heart Failure in Congenital Heart Disease: the role of myocardial fibrosis" (eIRB # 3665) including meeting all inclusion for that study (Aged 18-80, Known congenital heart disease).
4. Tetralogy of Fallot, cyanotic congenital heart disease, or a systemic right ventricle.

Exclusion Criteria:

1. Patient currently taking spironolactone or previously taking spironolactone within the last 6 months.
2. Serum potassium ≥5.0 mmol/L at the initial visit, if not taking potassium supplements. Patients will be eligible if a repeat potassium is <5.0 mmol/L after potassium supplements have been discontinued.
3. Moderate/severe systemic atrioventricular valve regurgitation,
4. Likely to undergo cardiac surgery, pacemaker implantation, or possible transplantation within one year (all self-reported),
5. Unwilling to commit to return visits including mandatory blood draws for potassium,
6. Renal insufficiency (estimated creatinine clearance < 30 ml/min/1.73m2),
7. Positive urine pregnancy test.
8. Any contraindication to MRI.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2016-06 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Broberg, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited at time of presentation for larger study. However, most did not meet enrollment criteria and could not be randomized.
Period: Overall Study
Arm/Group | Placebo | Spironolactone
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Spironolactone | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (6) | 38 (16) | 37 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Extracellular Volume Fraction
Description: extracellular volume fraction measured by T1 mapping with MRI
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: percentage of myocardium
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 8 | 7
percentage of myocardium | 30.1 (3.8) | 25.3 (1.5)

2. Secondary Outcome: 6-minute Walk Distance
Description: distance walked recorded in meters after 6 minutes on flat ground
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 8 | 7
meters | 516 (124) | 492 (138)

3. Secondary Outcome: Procollagen 3 NT Peptide
Time Frame: 12 months
Population: Limited samples obtained from participants
Measure: Mean (Standard Deviation); unit: mcg/l
Arm/Group | Placebo | Spironolactone
Number analyzed (Participants) | 1 | 3
mcg/l | 3 (.7) | 4.8 (1.2)

ADVERSE EVENTS:
Arm/Group | Placebo | Spironolactone
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No